CLINICAL TRIAL: NCT01413087
Title: A Multi-Center, Open-Label, Randomized, Phase 2b Study to Evaluate the Efficacy and Safety of BC-819 and Gemcitabine in Patients With Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Efficacy and Safety of BC-819 and Gemcitabine in Patients With Locally Advanced Pancreatic Adenocarcinoma
Acronym: LAPC-BC-819
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to Sponsor's decision, only 12 patients were randomized & completed study.
Sponsor: Anchiano Therapeutics Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-PAN-02
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Pancreas, Adenocarcinoma
Keywords: Pancreatic cancer; Gemcitabine; BC-819; Adenocarcinoma; Resectable; H19 gene; DTA-H19; BioCancell; inodiftagene vixteplasmid
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms | interventions — Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8 mg BC-819 and Gemcitabine (Experimental): gemcitabine dose of 1000mg/m2 + 8 mg of BC-819
  Interventions: Biological: Biological/Vaccine: BC-819
- 12 mg BC-819 and Gemcitabine (Experimental): gemcitabine dose of 1000mg/m2 + 12 mg of BC-819
  Interventions: Biological: Biological/Vaccine: BC-819

INTERVENTIONS:
Biological: Biological/Vaccine: BC-819 — Post screening and prior to randomization, all patients will receive gemcitabine by IV infusion at a dose of 1000mg/m2 once weekly for four weeks. They may also enter the study if they received up to 4 doses of gemcitabine before entering the study. In this case, they will be randomized immediately provided there is no evidence of disease progression.
  After randomization patients will receive 6 weekly IV infusions of gemcitabine at a dose of 1000mg/m2 + 7 intratumoral injections of BC-819 (8 mg or 12 mg according to allocations by randomization)
  Other Names: DTA-H19; inodiftagene vixteplasmid

SUMMARY:
This is a multicenter, open label, randomized, phase 2b study, designed to evaluate the safety and efficacy of patients with locally advanced pancreatic adenocarcinoma following intratumoral administration of BC-819 and intravenously administered gemcitabine. Intratumoral injections of BC-819 will be performed using endoscopic ultrasound (EUS).

Primary Objective: To assess the effect of intratumoral endoscopic ultrasound injection of BC-819 administered with intravenous gemcitabine on progression-free survival.

Secondary Objectives: To compare the effects of intratumoral injection of BC-819 administered in combination with intravenous gemcitabine vs. intravenous gemcitabine alone on:

Overall survival, Response rate, Resectability of the target tumor lesion, Quality of life, Safety, Serological Tumor Marker: CA 19-9, Duration of response, Failure-free survival

DETAILED DESCRIPTION:
BC-819 (also known as DTA-H19) is a double-stranded DNA plasmid, 4,560 base pairs (bp) in length, carrying the gene for the Diphtheria toxin A (DT-A) chain under the regulation of the H19 promoter. This is a Targeted Cancer Therapy; DT-A chain expression is triggered by the presence of H19 transcription factors that are only up-regulated in tumor cells. The selective initiation of toxin expression results in selective tumor cell destruction via inhibition of protein synthesis selectively in the tumor cell, enabling highly targeted cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females > 18 years of age
2. If female, must not be pregnant or nursing; women of child-bearing potential must practice a medically approved method of contraception
3. If male, must practice a medically approved method of contraception if have a partner of childbearing potential
4. Histologically or cytologically confirmed adenocarcinoma of the exocrine pancreas
5. Locally advanced pancreatic cancer (LAPC) that is clinically unresectable as defined in the NCCN Guidelines
6. Karnofsky performance status (KPS) ≥ 70% at baseline
7. Adequate hematological, renal, and hepatic function

   * Platelet count ≥ 100,000/mm3
   * Absolute neutrophil count (ANC) ≥ 1500/mm3
   * Hemoglobin ≥ 10.0 g/dL (may be achieved by transfusion)
   * Creatinine (≤ 1.5 x ULN)
   * ALT, AST (≤ 1.5 x ULN)
   * Total Bilirubin (≤ 1.5 x ULN)
8. Have a target tumor lesion in the pancreas ≤ 6 cm in diameter that is accessible for intratumoral administration by EUS guidance as determined by the physician performing the EUS injection
9. Have a biopsy specimen that is positive for H19 expression (grade 2 or greater staining determined by a pathologist). H19 expression can be determined based on a biopsy specimen collected before study participation, if available.
10. No prior diagnosis of malignancy within 3 years except for curatively treated non-melanoma skin or in situ malignancies
11. Able to comply with the protocol procedures
12. Able and willing to provide written (signed) Informed Consent to participate in the study

Exclusion Criteria:

1. Have distant metastatic spread (such as liver or lung metastases), peritoneal spread or malignant ascites. Regional lymph node involvement may be considered in accordance with the PI's judgment
2. Received any prior therapy for the treatment of pancreatic malignancy (including chemotherapy, immunotherapy, vaccines, monoclonal antibodies, major surgery, or irradiation, whether conventional or investigational, other than up to4 single doses of gemcitabine chemotherapy.Patients who received prior gemcitabine will only be eligible, if they enter the study without evidence of disease progression.
3. Known human immunodeficiency virus (HIV) or hepatitis C virus (HCV) or hepatitis B virus (HBV) infection
4. Have clinically significant pancreatitis within 12 weeks of treatment
5. Have a clinical history of significant coagulopathy
6. Have a medical condition contraindicated for endoscopic-guided delivery and/or for IV administration of Gemcitabine or any intercurrent medical illness or other medical condition that would in the judgment of the investigator compromise patient safety or the objectives of the study
7. Have participated in any experimental therapeutic research study with an unapproved drug within 4 weeks of the screening visit
8. Patients who require ongoing anticoagulation for pre-existing conditions, e.g., thrombophlebitis, pulmonary embolus or atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Winthrop University Hospital, Mineola, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
- Israel (6):
  - Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galil Maaravi, Nahariya
  - Tel Aviv Medical Center, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- 8 mg BC-819 and Gemcitabine: gemcitabine dose of 1000mg/m2 + 8 mg of BC-819
  Biological/Vaccine: BC-819: Post screening and prior to randomization, all patients will receive gemcitabine by IV infusion at a dose of 1000mg/m2 once weekly for four weeks. They may also enter the study if they received up to 4 doses of gemcitabine before entering the study. In this case, they will be randomized immediately provided there is no evidence of disease progression.
  After randomization patients will receive 6 weekly IV infusions of gemcitabine at a dose of 1000mg/m2 + 7 intratumoral injections of 8 mg BC-819
- 12 mg BC-819 and Gemcitabine: gemcitabine dose of 1000mg/m2 + 12 mg of BC-819
  Biological/Vaccine: BC-819: Post screening and prior to randomization, all patients will receive gemcitabine by IV infusion at a dose of 1000mg/m2 once weekly for four weeks. They may also enter the study if they received up to 4 doses of gemcitabine before entering the study. In this case, they will be randomized immediately provided there is no evidence of disease progression.
  After randomization patients will receive 6 weekly IV infusions of gemcitabine at a dose of 1000mg/m2 + 7 intratumoral injections of 12 mg BC-819
Period: Overall Study
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 8 mg BC-819 and Gemcitabine: gemcitabine dose of 1000mg/m2 + 8 mg of BC-819
  Biological/Vaccine: BC-819: Post screening and prior to randomization, all patients will receive gemcitabine by IV infusion at a dose of 1000mg/m2 once weekly for four weeks. They may also enter the study if they received up to 4 doses of gemcitabine before entering the study. In this case, they will be randomized immediately provided there is no evidence of disease progression.
  After randomization patients will receive gemcitabine at a dose of 1000mg/m2 + 7 intratumoral injections of 8 mg BC-819
- 12 mg BC-819 and Gemcitabine: gemcitabine dose of 1000mg/m2 + 12 mg of BC-819
  Biological/Vaccine: BC-819: Post screening and prior to randomization, all patients will receive gemcitabine by IV infusion at a dose of 1000mg/m2 once weekly for four weeks. They may also enter the study if they received up to 4 doses of gemcitabine before entering the study. In this case, they will be randomized immediately provided there is no evidence of disease progression.
  After randomization patients will receive gemcitabine at a dose of 1000mg/m2 + 7 intratumoral injections of 12 mg BC-819
- Total: Total of all reporting groups
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (6.7) | 62.2 (13.0) | 67.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: To compare the effect of intratumoral endoscopic ultrasound injection of BC-819 administered with intravenous gemcitabine on progression-free survival. PFS was defined as the time from the date of consent until objective tumor progression or death. Median PFS by Kaplan-Meier analysis was used for evaluation. The target tumor lesion was identified and the longest diameter of the target lesion was measured according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines. For disease evaluations after treatment, scans conducted at baseline that were used for tumor measurements were repeated.
Time Frame: 24 months
Population: ITT comprised of all subjects who received any treatment with either gemcitabine or BC-819 and whose tumors were positive for H19. All 12 patients were included in the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
months | 9.3 [2.6 to 26.3] | 7.6 [6.3 to 10.7]
Statistical Analysis 1: Comparison: 8 mg BC-819 and Gemcitabine vs 12 mg BC-819 and Gemcitabine; Test type: Superiority; p = 0.483, Log Rank; P value by log-rank test for the difference between treatment groups

2. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated from the date of consent until death due to any cause.
Time Frame: 24 months
Population: ITT population comprised all subjects who received any treatment with either gemcitabine or BC-819 and whose tumors were positive for H19. All 12 patients were included in the ITT population
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
years | 9.9 [5.4 to 26.4] | 8.5 [6.8 to NA] — Upper limit of OS not reached
Statistical Analysis 1: Comparison: 8 mg BC-819 and Gemcitabine vs 12 mg BC-819 and Gemcitabine; Test type: Superiority; p = 0.992, Log Rank; P value by log-rank test for the difference between treatment groups

3. Secondary Outcome: Response Rate of Target Lesion
Description: Response rate will be assessed both for the primary target tumor lesion alone and overall, including development of metastases. Target tumor lesions are identified and the longest diameter of the target lesion is measured by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines.
  Complete response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also show an increase of at least 5 mm.
  Stable Disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 8 weeks
Population: ITT population comprised of all subjects who received any treatment with either gemcitabine or BC-819 and whose tumors were positive for H19. All 12 patients were included in the ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
Participants
  Complete Response | 0 | 0
  Partial Response | 1 | 0
  Stable Disease | 2 | 6
  Progressive Disease | 1 | 0
  Inevaluable - Missing Postbaseline Scan | 2 | 0

4. Secondary Outcome: Resectability of the Target Tumor Lesion
Description: Resectability of the target tumor lesion was determined by CT/MRI as defined in the National Comprehensive Cancer network (NCCN) guidelines. Resectable tumors have no arterial tumor contact (celiac axis [CA], superior mesenteric artery [SMA], or common hepatic artery [CHA]) and no tumor contact with the superior mesenteric vein (SMV) or portal vein (PV) or ≤180° contact without vein contour irregularity. *Not Applicable refers to another clinically significant abnormality that interfered with resectability determination of the target tumor lesion.
Time Frame: an average of 16 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
Participants
  Not Resectable | 5 | 6
  Not Applicable* | 1 | 0

5. Secondary Outcome: Quality of Life (QoL) Assessed by Karnofsky Performance Status (KPS)
Description: Quality of life will be assessed by the The Karnofsky Performance Status (KPS) Index. KPS scores over time will be compared to those at baseline and changes from baseline will be presented.
  KPS scores are on a scale (0, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100) of 0 (dead) to 100 (Normal no complaints; no evidence of disease).
Time Frame: Screening, Visit 4 (post gemcitabine induction), Visit 9 (5 weeks), Visit 13 (9 weeks)
Population: as for outcome 3
Measure: Median (Full Range); unit: score on a scale
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
score on a scale
  Screening | 90 [80 to 100] | 90 [80 to 100]
  Visit 4 (pre-randomization) | 90 [90 to 90] | 85 [80 to 100]
  Visit 9 (Week 5) | 80 [80 to 90] | 90 [80 to 90]
  Visit 13 (Week 9) | 80 [80 to 90] | 90 [80 to 90]

6. Secondary Outcome: Quality of Life Using the Functional Assessment of Cancer Therapy-General (FACT-G) Questionnaire
Description: The FACT-G is a 27-item compilation of general questions divided into 4 primary QoL domains: physical well-being, social/family well-being, emotional well-being and functional well-being. The total FACT-G scores will be summarized by descriptive statistics (e.g., n, mean, median, standard deviation and range). The individual FACT-G score will be presented by frequency and percentage. Scores range from 0-108. High total scores represent better general QoL.
Time Frame: Screening, Visit 4 (post gemcitabine induction), Visit 9 (5 weeks), Visit 13 (9 weeks), every 6 months after Visit 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
units on a scale
  Screening | 71.8 (11.8) | 81.9 (14.0)
  Max change from baseline | -1.3 (18.5) | -2.5 (18.8)

7. Secondary Outcome: Serological Tumor Marker: CA 19-9
Description: Serum was collected for quantitative measurement of CA 19-9.
Time Frame: 24 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
U/mL
  Screening | 1025.9 (1090.6) | 587.7 (340.1)
  Nadir value | 369.8 (511.7) | 149.1 (97.0)
  Change at Nadir | -656.1 (887.7) | -438.6 (252.2)

8. Secondary Outcome: Extent of Exposure - Gemcitabine Total Exposure (g)
Description: Measured by the average and median number of exposure of the patients to BC-819 and gemcitabine.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
g | 20.1 (9.5) | 21.3 (11.9)

9. Secondary Outcome: Extent of Exposure - Gemcitabine Total Number of Treatments
Description: Measured by the average and median number of treatments of the patients to BC-819 and gemcitabine.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of treatments
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
number of treatments | 17.3 (14.9) | 15.3 (12.7)

10. Secondary Outcome: Extent of Exposure - BC-819 Total Exposure (mg)
Description: Measured by the average and median exposure of the patients to BC-819 and gemcitabine.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
mg | 68.0 (29.8) | 118.0 (41.2)

11. Secondary Outcome: Extent of Exposure - BC-819 Total Number of Treatments
Description: Measured by the average and median number of treatments of the patients to BC-819 and gemcitabine.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of treatments
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
Number analyzed (Participants) | 6 | 6
number of treatments | 10.7 (8.4) | 11.2 (6.0)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse Events were only assessed after randomization to either dose level of BC-819.
Groups:
- 8 mg BC-819 and Gemcitabine: gemcitabine dose of 1000mg/m2 + 7 intratumoral injections of 8 mg BC-819
  Biological/Vaccine: BC-819: Post screening and prior to randomization, all patients will receive gemcitabine by IV infusion at a dose of 1000mg/m2 once weekly for four weeks. They may also enter the study if they received up to 4 doses of gemcitabine before entering the study. In this case, they will be randomized immediately provided there is no evidence of disease progression.
  After randomization patients will receive gemcitabine at a dose of 1000mg/m2 + 7 intratumoral injections of 8 mg BC-819
- 12 mg BC-819 and Gemcitabine: gemcitabine dose of 1000mg/m2 + 7 intratumoral injections of 12 mg BC-819
  Biological/Vaccine: BC-819: Post screening and prior to randomization, all patients will receive gemcitabine by IV infusion at a dose of 1000mg/m2 once weekly for four weeks. They may also enter the study if they received up to 4 doses of gemcitabine before entering the study. In this case, they will be randomized immediately provided there is no evidence of disease progression.
  After randomization patients will receive gemcitabine at a dose of 1000mg/m2 + 7 intratumoral injections of 12 mg BC-819
Arm/Group | 8 mg BC-819 and Gemcitabine | 12 mg BC-819 and Gemcitabine
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/6
Serious Adverse Events (participants affected / at risk) | 5/6 | 5/6
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg BC-819 and Gemcitabine (N=6) | 12 mg BC-819 and Gemcitabine (N=6)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Generalized Edema (General disorders) | 1 (1) | 0 (0) — Subjects with SAEs related to gemcitabine with reasonable possibility
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Reasonable possibility of relationship to study procedure.
Frequent bowel movement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 2 (3) — One subject who reported this SAE had a reasonable possibility of relationship to study procedure
Duodenitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stent malfunction (Product Issues) | 0 (0) | 1 (2) — Reasonable possibility of relationship to study procedure.
Melena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Bilateral pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Injection site abscess (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Reasonable possibility of relationship to study procedure.
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg BC-819 and Gemcitabine (N=6) | 12 mg BC-819 and Gemcitabine (N=6)
Nausea (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 4 | 1
Asthenia (General disorders) | 2 | 1
Peripheral edema (Eye disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 1
Increased blood bilirubin (Investigations) | 0 | 3
Increased gamma glatamyl transferase (Investigations) | 1 | 2
Decreased neutrophil count (Investigations) | 1 | 2
Increased alanine aminotransferase (Investigations) | 0 | 2
Increased aspartate aminotransferase (Investigations) | 0 | 2
Increased blood alkaline phosphatase (Investigations) | 0 | 2
Decreased haemoglobin (Investigations) | 1 | 1
Abnormal liver function tests (Investigations) | 1 | 1
Decreased platelet count (Investigations) | 1 | 1
Decreased weight (Investigations) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 2
Chills (General disorders) | 1 | 0 (0) — Subjects with AEs Related to BC-819 with reasonable possibility
Nausea (Gastrointestinal disorders) | 3 | 3 — Subjects with AEs Related to gemcitabine with reasonable possibility
Vomiting (Gastrointestinal disorders) | 2 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility
Fatigue (General disorders) | 1 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility
Anemia (Blood and lymphatic system disorders) | 1 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility
Constipation (Gastrointestinal disorders) | 1 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility
Diahrrea (Gastrointestinal disorders) | 1 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility
Asthenia (General disorders) | 1 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 — Subjects with AEs Related to gemcitabine with reasonable possibility
Stomatitis (Gastrointestinal disorders) | 1 | 0 — Subjects with AEs Related to gemcitabine with reasonable possibility
Peripheral edema (General disorders) | 1 | 0 — Subjects with AEs Related to gemcitabine with reasonable possibility
Cellulitis (Infections and infestations) | 1 | 0 — Subjects with AEs Related to gemcitabine with reasonable possibility
Abnormal liver function test (Investigations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 — Subjects with AEs Related to gemcitabine with reasonable possibility
Decreased platelet count (Blood and lymphatic system disorders) | 0 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility
Decreased weight (Investigations) | 0 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 — Subjects with AEs Related to gemcitabine with reasonable possibility
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 — Subjects with AEs Related to gemcitabine with reasonable possibility

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days